CLINICAL TRIAL: NCT06274203
Title: Safety and Efficacy of Monthly High-Dose Vitamin D3 Supplementation in Children and Adolescents With Sickle Cell Disease and Healthy Counter Parents
Brief Title: High Dose Vitamin D Supplementation in Children With Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Diana Hanna Abdelmalek Hanna, Lecturer of pediatric hematology and oncology, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10584-2/5-2023
Record Dates: First submitted 2024-02-13; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Sickle Cell Disease; Vitamin D Deficiency; Health Related Quality of Life; Hand Grip Strength; Bone Mineral Density
MeSH Terms: conditions — Anemia, Sickle Cell; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral vitamin D3 (Experimental): Monthly oral vitamin D3 dose (100,000 IU,150,000 IU, and 200,000 IU)
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — Subjects within SCD as well as healthy controls, received monthly oral vitamin D3 dose, for 6 months, according to the baseline status of vitamin D as follows: sufficient (>30 ng/mL): 100,000 IU, insufficient (20-29.9 ng/mL): 150,000 IU, and deficient (<20 ng/mL): 200,000 IU.

SUMMARY:
Suboptimal vitamin D status is well reported in sickle cell disease (SCD) patients and associated with a negative impact on health-related quality of life (HRQL). The investigators enrolled 42 SCD patients and 42 healthy controls, subjects within each group received monthly oral vitamin D3 dose according to the baseline status of vitamin D as follows: sufficient: 100,000 IU, insufficient: 150,000 IU, and deficient: 200,000 IU. The investigators assessed safety and efficacy on normalization of vitamin D level, bone mineral density (BMD), hand grip strength (HGS), and HRQL.

ELIGIBILITY:
Inclusion Criteria:

* children with SCD (HbSS, hemoglobin sickle beta zero (HbSβ0) thalassemia genotype), aged ≤ 18 years old, male or female study participants who were at a steady state (≥ one month from blood transfusion and ≥ 14 days from any acute sickle complication as hospitalization for Vaso occlusive crisis (VOC) or acute chest syndrome (ACS)), stable Hb level near their usual baseline and stable dose of Hydroxyurea (HÚ) mg/kg for at least 90 days prior to enrollment.
* A control group of 42 healthy age and sex-matching children

Exclusion Criteria:

* SCD patients who are on chronic blood transfusion therapy
* Comorbid chronic conditions
* Use of medications known to interfere with calcium or vitamin D absorption or metabolism
* Known hypercalcemia or vitamin D hypersensitivity
* Use of vitamin D therapy to treat vitamin D deficiency or rickets
* Urolithiasis, liver or renal impairment, and malabsorption disorders.
* Obese children with body mass index (BMI) > 85th percentile for age and sex

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Serum 25(OH)D level | up to 6 months
  Serum 25(OH)D level change from baseline at 6 months

SECONDARY OUTCOMES:
Bone mineral density (BMD) | up to 6 months
  BMD was evaluated at the posterior-anterior spine, Z-scores were used to interpret the results, with Z-scores less than -2 standard deviation (SD) being regarded as abnormal
Maximum handgrip strength (HGS) | up to 6 months
  Hand grip power using a handheld dynamometer.
Health related quality of life (HRQL) | up to 6 months
  Health related quality of life (HRQL) assessed by HRQL questionnaires, The questionnaire was divided into eight subscales: physical function, role limitations resulting from physical health, bodily pain, general health perception, vitality, social function, role limitations resulting from emotional problems, and mental health. For each subscale: higher score indicated good health and ranged from 0 to 100.
Serum concentrations of C reactive protein (CRP) | up to 6 months
  Serum concentrations of inflammatory marker (CRP) level change from baseline
Serum concentrations of Erythrocyte sedimentation rate (ESR) | up to 6 months
  Serum concentrations of inflammatory marker (ESR) level change from baseline
Safety reporting of any adverse events | up to 6 months
  e.g. nausea, drowsiness, vomiting, loss of appetite, constipation, confusion, cardiac arrhythmias, renal failure, coma
Safety measurements of serum Ca | at 3 and 6 months
  serum Ca levels
childhood health assessment | up to 6 months
  Assessed by childhood health assessment questionnaire (CHAQ), There are four potential responses to each question: "without any difficulty" (score 0); "with some difficulty" (score 1); "with much difficulty" (score 2); and "unable to do" (score 3). A summary score known as CHAQ-DI/, which varies from 0 to 3, is calculated by averaging the highest score in each domain. For a CHAQ-DI score to be considered minimally clinically significant, it must be ≥ 0.75.
Safety measurements of serum 25(OH)D levels | at 3 and 6 months
  serum 25(OH)D levels

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig university, Zagazig, Sharqia Province, Egypt

REFERENCES:
- [Derived] Hanna D, Kamal DE, Fawzy HM, Abd Elkhalek R. Safety and efficacy of monthly high-dose vitamin D3 supplementation in children and adolescents with sickle cell disease. Eur J Pediatr. 2024 Aug;183(8):3347-3357. doi: 10.1007/s00431-024-05572-w. Epub 2024 May 14. PMID 38743288